CLINICAL TRIAL: NCT00240786
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating Acetaminophen Extended Release (1950 mg/Day or 3900 mg/Day) in the Treatment of Osteoarthritis of the Hip or Knee
Brief Title: An Effectiveness and Safety Study of Two Doses of Acetaminophen Extended Release Caplets in the Treatment of Osteoarthritis of the Hip or Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002485
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis hip; osteoarthritis knee; acetaminophen
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee

INTERVENTIONS:
Drug: acetaminophen extended release

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of 650 mg and 1300 mg acetaminophen extended release given three times a day for the relief of signs and symptoms of osteoarthritis of the hip or knee for a period of 12 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to determine the safety and effectiveness of 650 mg and 1300 mg acetaminophen extended release given three times a day as compared with placebo, for the relief of signs and symptoms of osteoarthritis of the hip or knee for a period of 12 weeks. Propoxyphene Hydrochloride capsules 65 mg are used as rescue medication if subjects experience inadequate pain relief. The primary efficacy assessments are the average change from baseline to the final on-therapy visit for the WOMAN pain subscale score and the WOMAC physical function subscale scare, and the subject's average global assessment of their response to therapy through the final on-therapy visit. Safety assessments at study visits consist of monitoring adverse events, vital signs, study joint assessments and clinical laboratory determinations. The hypothesis is that 1950 mg per day and/or 3900 mg per day acetaminophen extended release are superior to placebo for the relief of the signs and symptoms of osteoarthritis of the hip or knee with respect to all three primary efficacy endpoints. Treatment consisted of either one 650 mg acetaminophen extended release caplet plus one placebo caplet (acetaminophen 1950 mg group); two 650 mg acetaminophen extended release caplets (acetaminophen 3900 mg group); or two placebo caplets administered orally every eight hours for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptomats of osteoarthritis of the hip or knee for a minimum of six months
* History of hip or knee pain due to osteoarthritis requiring the use of NSAIDs, acetaminophen, or another analgesic agent on a regular basis (>= three days per week) for at least three months before the screening visit
* History of positive therapeutic benefit with acetaminophen use for osteoarthritis pain
* History of osteoarthritis pain (moderate, moderately severe, or severe) of the hip or knee when not taking osteoarthritis analgesic medication
* Must have a pain level of moderate or moderately severe for 24 hours over the previous 24 hours prior to the baseline visit, and at baseline, demonstrate a 20% or greater increase in the pain subscale score, relative to the score at screening

Exclusion Criteria:

* History of surgery, including arthroscopy, or major trauma to the study joint in the previous six months before the screening visit
* Grade 1 or grade 4 severity of the study joint based on the Kellgren and Lawrence radiographic criteria
* Maximum osteoarthritis pain intensity of none, mild or severe experienced over the previous 24 hours of the baseline visit
* Signs of clinically important active inflammation of the study knee joint including redness, warmth and/or a large, bulging effusion with the loss of normal contour at the screening and/or baseline visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2002-04; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Average change from baseline to the final on-therapy visit for - WOMAC pain subscale score; WOMAC physical function subscale score; and subject's average global assessment of response to therapy through the final on-therapy visit

SECONDARY OUTCOMES:
Average change from baseline to final on-therapy visit for WOMAC stiffness subscale score; average change from baseline to final on-therapy visit for total WOMAC Index; average number of propoxyphene HCl rescue medication capsules per day while in study

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Kuffner EK, Temple AR, Cooper KM, Baggish JS, Parenti DL. Retrospective analysis of transient elevations in alanine aminotransferase during long-term treatment with acetaminophen in osteoarthritis clinical trials. Curr Med Res Opin. 2006 Nov;22(11):2137-48. doi: 10.1185/030079906x148346. PMID 17076974
- See also: An Effectiveness and Safety Study of Two Doses of Acetaminophen Extended Release Caplets in the Treatment of Osteoarthritis of the Hip or Knee — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=902&filename=CR002485_CSR.pdf